CLINICAL TRIAL: NCT01608750
Title: The Efficacy of Pantoprazole Treatment in Patients With Functional Dyspepsia: Randomised, Double-blind, Placebo-controlled Trial.
Brief Title: The Efficacy of Pantoprazole Treatment in Patients With Functional Dyspepsia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Birol Baysal, Gastroenterologist, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B.30.2.BAV.0.05.05/331
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Nonulcer Dyspepsia
MeSH Terms: interventions — Pantoprazole; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pantoprazole (Experimental)
  Interventions: Drug: Pantoprazol
- folic acid (Placebo Comparator)
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Pantoprazol — 40mg/day, oral, 28 days
  Arms: pantoprazole
Drug: Folic Acid — 5 mg/day, oral, 28 days
  Arms: folic acid

SUMMARY:
The aim of our study is to evaluate the effectiveness of proton pump inhibitor (PPI) treatment in patients with functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years with symptoms of dyspepsia,
* no evidence of organic disease.

Exclusion Criteria:

* Patients with alarm symptoms,
* Severe concomitant illness,
* Pregnancy or lactation,
* Alcohol or drug abuse,
* Use of aspirin or other non-steroidal anti-inflammatory drugs antibiotics, H2 receptor blockers, bismuth, or proton pump inhibitors in the preceding two weeks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of pantoprazole treatment in patients with functional dyspepsia measured by symptoms scale. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem medical faculty, Istanbul, Turkey (Türkiye)